CLINICAL TRIAL: NCT07241221
Title: Antenatal Myo-inositol Supplementation in Pre-existing Diabetes to Promote Normal Neonatal Outcomes
Brief Title: Antenatal Myo-inositol Supplementation in Pre-existing Diabetes
Acronym: AMulet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2024-4610
Record Dates: First submitted 2025-09-18; First posted 2025-11-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Perinatal and Neonatal Outcomes in Pregnancies With Type 2 Diabetes Mellitus (T2DM)
Keywords: Diabetes; Pregnancy; Myo-inositol; Folic acid; Dietary Supplement; Birthweight; Prematurity; Neonatal Intensive Care Unit Admission; Stillbirth; Neonatal Death; Neonatal Complications; Maternity Complications
MeSH Terms: conditions — Diabetes Mellitus; Birth Weight; Premature Birth; Stillbirth; Perinatal Death | interventions — Inositol

STUDY DESIGN:
Intervention Model Description: Two parallel arm, double-blinded, placebo-controlled, randomized controlled trial design in a 1:1 ratio. Pregnant women with T2DM will be randomly assigned to either the intervention group (receiving supplementation of myo-inositol with folic acid) or the control group (receiving supplementation with folic acid only). Randomization will be stratified by ethnicity to ensure a balanced allocation between arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (myo-inositol and folic acid supplement) (Experimental): Participants in the intervention arm will receive a total of 4 g/day of myo-inositol and 300 mcg/day of folic acid, divided into two daily doses.
  Interventions: Dietary Supplement: Myo-inositol and folic acid supplement
- Control (folic acid supplement) (Active Comparator): Participants in the control arm will receive a total of 300 mcg/day of folic acid, divided into two daily doses.
  Interventions: Dietary Supplement: Folic acid supplement

INTERVENTIONS:
Dietary Supplement: Myo-inositol and folic acid supplement — Participants will take 4 capsules in the morning and 4 capsules in the evening, each capsule containing 500 mg of myo-inositol and 37.5 mcg of folic acid. Capsules are to be swallowed whole with a drink, starting from 12-16 weeks' gestation and continued until delivery.
  Arms: Intervention (myo-inositol and folic acid supplement)
Dietary Supplement: Folic acid supplement — Participants will take 4 capsules in the morning and 4 capsules in the evening, each capsule containing 37.5 mcg of folic acid. Capsules are to be swallowed whole with a drink, starting from 12-16 weeks' gestation and continued until delivery.
  Arms: Control (folic acid supplement)

SUMMARY:
This feasibility pilot study aims to gather data that can guide the design of a larger, more comprehensive trial to establish the effects of myo-inositol supplementation on supporting healthy outcomes in pregnancies complicated by Type 2 Diabetes Mellitus (T2DM). It seeks to assess myo-inositol's potential to support fetal and neonatal health, and optimise maternity outcomes as a complementary approach and adjuvant to existing diabetes mellitus therapies, as well as investigate the underlying biological mechanisms.

DETAILED DESCRIPTION:
The "Antenatal Myo-inositol supplementation in pre-existing diabetes to promote normal neonatal outcomes (AMulet)" pilot study aims to inform the design of a future double-blind randomised controlled trial which can assess the benefits of myo-inositol supplementation in pregnant women with T2DM. Despite provision of the international standard of care, pregnancies complicated by diabetes remain at high risk of adverse perinatal and neonatal outcomes. Offspring exposed to maternal diabetes in-utero also face increased risks of obesity and cardiometabolic diseases later in life. Myo-inositol supplementation has been trialled in pregnancy for the prevention and treatment of gestational diabetes, as well as in non-pregnant adults with T2DM, where improvements in glycaemic regulation and reduced insulin resistance have been observed with supplementation. However, myo-inositol supplementation has not yet been studied in pregnancies with T2DM. The primary aim of the AMulet trial would be to assess whether myo-inositol supplementation in pregnancies with T2DM can support normal fetal size and neonatal wellbeing. The present AMulet pilot study will assess the feasibility and acceptability of conducting such a trial and, additionally, seek to investigate the biological mechanisms through which myo-inositol may influence maternal and offspring health outcomes.

This pilot will recruit 182 pregnant women with T2DM between 12-16 weeks' gestation into a double-blind placebo-controlled randomized study. All participants will be randomly assigned to either an intervention group (receiving supplementation of myo-inositol with folic acid) or a control group (receiving supplementation with folic acid only). Supplementation will be in the form of similar looking capsules to be taken twice daily from recruitment until delivery.

Data and samples will be collected longitudinally across three study visits during pregnancy that will be arranged to coincide with routine antenatal clinic visits where possible, and a fourth visit soon after delivery. Additionally, there will be two re-supply visits and a post-delivery videoconference call. Other study data comprising antenatal, peripartum, fetal and neonatal outcomes will be extracted from medical records during pregnancy and post-delivery to assess the primary and secondary outcomes.

The binary composite primary outcome of normal fetal/neonatal size and wellbeing will be assessed by analyses on an intention-to-treat basis. Secondary outcomes, comprising maternity and other infant outcomes, will be assessed and quantified in terms of relative risk or mean differences between study groups. Adverse events, participant feedback as well as mechanistic understanding will be obtained.

This structured approach will inform the design of a future RCT by gathering data on feasibility and acceptability, identifying potential issues in protocols and data collection tools, and facilitating sample size calculations for the main trial which will aim to support the optimization of maternal and offspring health outcomes in pregnancies complicated by pre-existing T2DM.

ELIGIBILITY:
Inclusion Criteria

* Pregnant women aged 21 years to 45 years old at the time of recruitment
* Ongoing, viable, singleton intrauterine pregnancy
* Between 12+0 days-16+6 days weeks' gestation at recruitment
* T2DM diagnosed by a documented 75g Oral Glucose Tolerance Test (OGTT) showing a fasting glucose of >7 mmol/L or 2h glucose >11.1 mmol/L, or an HbA1C >6.5%, either prior to pregnancy or during the first 16 weeks of the index pregnancy
* Intend to receive antenatal care and give birth at NUH
* Willing to provide written, informed consent
* Able to swallow capsules and comply with trial procedures

Exclusion Criteria

* Known or suspected fetal aneuploidy or genetic/structural anomaly
* Severe allergy to food items requiring carriage of an Epipen at all times

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite of fetal/neonatal wellbeing | From birth until 4 weeks post-delivery
  Number and proportion of cases displaying all of the following outcomes of (1) being appropriately-grown-for-gestational-age (AGA; 10th-90th centile in weight) at birth; (2) delivered at term (37 weeks+0 days gestation or more); (3) no admission to the neonatal unit in the first 4 weeks of life; and (4) alive at delivery and at 4 weeks post-delivery. Results will also be presented as a relative risk with 95% confidence intervals, with and without adjustment for important covariates, as well as with and without stratification for baseline HbA1C (high/low), pre-pregnancy insulin treatment, duration since T2DM diagnosis (<1y, >1y), and in per-protocol analyses.

SECONDARY OUTCOMES:
Intrauterine fetal growth and wellbeing as assessed by antenatal serial ultrasound scans | Up to 38 weeks duration, from the earliest scan in pregnancy ~5-6 weeks' gestation until delivery of the baby between 22-42 weeks' gestation.
  Mean differences in cross-sectional comparisons and longitudinal changes in measured biometric parameters, derived size/weight estimates and Doppler assessments, as well as differences in the velocity of growth, peak/nadir in the velocity of growth and its gestational timing, and the fastest/slowest change in growth velocity and its gestational timing, with and without adjustment for important covariates.
Neonatal anthropometry and body composition | Birth till 4-6 weeks post-delivery
  Number and proportion, and relative risks, of macrosomia (birthweight >4000 g), low birthweight (<2500 g), Large-for-Gestational-Age (LGA; birthweight >90th centile), and Small-for-Gestational-Age (SGA; birthweight <10th centile), and mean differences or categorically-defined outcomes of birthweight, birth length, head circumference, abdominal circumference, mid-arm circumference, skinfold thickness, fat mass, fat-free mass, and percentage body fat (assessed by air displacement plethysmography, PEAPOD), with and without adjustment for important covariates. Continuous data to be standardised to z-scores, where appropriate.
Other perinatal and neonatal outcomes | Birth till 4-6 weeks post-delivery
  Number and proportion, and relative risks, of neonatal respiratory distress (aetiology and treatment required), neonatal hypoglycemia, number of hypocount values <2.6 mmol/L, hyperbilirubinemia requiring phototherapy or exchange transfusion, neonatal sepsis (early and late onset, aetiology and treatment required), shoulder dystocia, birth trauma, hypoxic ischaemic encephalopathy/intracranial haemorrhage, neonatal unit admission, or stillbirth/neonatal death, as well as mean differences in the levels of glycaemia and bilirubinaemia, and in the duration of respiratory support, phototherapy and neonatal unit/hospital stay, with and without adjustment for important covariates. Continuous data to be standardised to z-scores, where appropriate.
Fetal (cord) insulinaemia and C-peptide | At birth
  Number and proportion, and relative risks of fetal hyperinsulinaemia or high C-peptide concentration, and mean difference in insulin or C-peptide concentrations in umbilical cord blood (where obtainable); with and without adjustment for important covariates
Maternal glycaemic control | Up to 100 weeks duration, from within a year before conception (last recorded before conception) or early pregnancy (between conception and recruitment between ~12-16 weeks gestation), until the delivery of the baby (between 22-42 weeks gestation).
  Mean differences and change in blood glucose levels (monitored through self-blood glucose monitoring or continuous glucose monitoring, CGM), other CGM parameters, markers of glycemic control, the frequency of participant-managed hypoglycemic episodes, proportional increases in metformin or insulin doses, and mean differences in daily insulin requirements per kilogram (kg) of body weight, proportion requiring other diabetes treatments, mean differences and change in HbA1C and HOMA-IR; with and without adjustment for important covariates. Continuous data to be standardised to z-scores, where appropriate.
Hypertensive disorders of pregnancy | Between time of recruitment (~12 to 16 weeks of gestation) and 4-6 weeks post-delivery
  Number and proportion, and relative risks, of pre-eclampsia/eclampsia, superimposed pre-eclampsia on chronic hypertension, and pregnancy-induced hypertension (as a composite and as individual complications), as well as difference in the gestational age of onset or diagnosis and severity of disorder, with and without adjustment for important covariates.
Gestational age at delivery and preterm prelabour rupture of membranes (PPROM) | Between time of recruitment (~12 to 16 weeks of gestation) and delivery
  Number and proportion, and relative risks, of PPROM and preterm delivery (spontaneous and/or iatrogenic births), reasons for preterm birth, as well as the gestational ages at delivery and at PPROM will be presented, with and without adjustment for important covariates.
Gestational weight gain | Up to 100 weeks duration; From pre-pregnancy (last recorded weight before conception) or earliest recorded weight in pregnancy (between conception and recruitment) to the last recorded weight before delivery (22-42 weeks gestation).
  Mean differences in the total weight a woman gains during pregnancy, measured in kilograms (kg), as well as the rate of weight gain over the second and third trimesters of pregnancy (kg/week). Proportional differences in the categorisation of weight gain by the Institute of Medicine (IOM) guidelines as insufficient, appropriate, or excessive (considering the mother's pre-pregnancy BMI), with and without adjustment for important covariates
Maternal depressive and anxiety symptoms | Between time of recruitment (~12 to 16 weeks of gestation) and 4-6 weeks post-delivery
  Mean differences and change from baseline in scores of maternal depression and anxiety symptoms on validated questionnaires (Edinburgh Postnatal Depression Scale and State-Trait Anxiety Inventory), and proportional differences between groups in those with higher and lower scores, with and without adjustment for important covariates. Continuous data to be standardised to z-scores, where appropriate.
Mode of delivery | At delivery
  Number and proportion, and relative risks, of caesarean section, primary caesarean section, emergency caesarean section, and instrumental delivery, with and without adjustment for important covariates.
Postpartum blood loss | At delivery and up to 4-6 weeks post-delivery
  Number and proportion, and relative risks, of major postpartum haemorrhage (primary and secondary), and mean differences in the volume of blood loss (primary and secondary), with and without adjustment for important covariates.
Other antenatal and peripartum events | From conception to 4-6 weeks post-delivery
  Number and proportion, and relative risks, of antenatal complications such as intrahepatic cholestasis, placental abruption and antepartum haemorrhage, and peripartum events encompassing type of onset/induction and progress of labour, requirement for labour augmentation, non-reassuring cardiotocography suggestive of fetal compromise, meconium-stained liquor, shoulder dystocia, perineal trauma, admission to high-dependency/intensive care unit, and other relevant complications, as well as mean differences in the duration of each stage of labour and entire labour, and length of maternal HDU/ICU/hospital stay, with and without adjustment for important covariates.
Circulating, urinary and placental inositol and inositol-metabolite concentrations | Between time of recruitment (~12 to 16 weeks of gestation) and delivery
  Mean differences in cross-sectional comparisons and longitudinal changes from baseline in maternal circulation and urinary concentrations of myo-inositol and the other 4 inositol isomers, and inositol metabolites, as well as mean differences in circulating fetal/cord concentrations of these inositols/inositol-metabolites at birth, and in placental and fetal membrane tissues; with and without adjustment for important covariates.
Multi-Omic Profiling | Between the time of recruitment (~12 to 16 weeks of gestation) and delivery
  Differences in the characteristics and quantities of each element/class of the biochemical, metabolic, metabolomic, hormonal, chemoadipocytokine, proteomic, lipidomic, genomic, epigenomic and transcriptomic profiles as well as tissue tensile strength (where applicable) in maternal blood & urine, fetal (umbilical cord) blood & tissue, placenta and fetal membranes.
Stool microbiota composition and activity | Between the time of recruitment (~12 to 16 weeks of gestation) and 4-6 weeks post-delivery
  Descriptive and quantifiable differences in metagenomics and metatranscriptomics, reflecting microbial diversity, the relative abundance of key bacterial species, and metabolic activity in maternal and neonatal stool. Continuous data to be standardised to z-scores, where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Shiao-Yng Chan, MBBChir (UK), FRCOG (UK), PhD, Principal Investigator — National University of Singapore, National University Hospital Singapore, Institute for Human Development and Potential (A*STAR)
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No